CLINICAL TRIAL: NCT03435445
Title: Use of Web as a Tool to Promote Weight Loss in Overweight and Obese Adults
Brief Title: Online Platform for Healthy Weight Loss (POEmaS)
Acronym: POEmaS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Collaborators: Ministry of Science and Technology, Brazil (Other)
Responsible Party: Principal Investigator, Antonio Luiz Pinho Ribeiro, Full Professor, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 73545717500005149
Record Dates: First submitted 2018-01-30; First posted 2018-02-19 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Obesity; Overweight
Keywords: obesity; overweight; telemedicine; ehealth
MeSH Terms: conditions — Obesity; Overweight | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: 3 arms: Experimental group 1 receives diet, physical change and behavior change recommendations via an online platform for 24 weeks; Experimental Group 2 receives recommendations via an online platform plus a dietitian coaching via the online platform for 24 weeks; Control groups receives a minimal intervention with access to diet and physical change recommendations videos. After 24 weeks, the control group will gain access to the online platform.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Online platform group (Experimental): Online platform with diet, physical activity and behavior change recommendations for 24 weeks
  Interventions: Behavioral: Online platform group
- Online dietitian coaching (Experimental): Diet, physical activity and behavior change recommendations for 24 weeks and online sessions with a dietitian specialist for 12 weeks
  Interventions: Behavioral: Online platform group; Behavioral: Online dietitian coaching
- Control group (Active Comparator): Videos with diet, physical activity and behavior change recommendations for 24 weeks
  Interventions: Behavioral: Control group

INTERVENTIONS:
Behavioral: Online platform group — The online platform has social network, gamification and short-text sessions.
  Arms: Online dietitian coaching; Online platform group
Behavioral: Online dietitian coaching — Dietitian coaching refers to individual online sessions between a dietitian and participants to strengthen dietary recommendations
  Arms: Online dietitian coaching
Behavioral: Control group — Minimal intervention with four videos with diet, physical activity and behavior change recommendations
  Arms: Control group

SUMMARY:
Clinical trial to test the efficacy of an online platform based on behavior change principles in promoting weight loss among overweight and obese students and employees of the Federal University of Minas Gerais. The hypothesis is that participants of the group which use the platform with or without a dietitian coaching will lose more weight than those allocated to the group who receives dietary and physical activity orientations by educational videos only.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index >=25 kg/m2
* intention to lose weight by healthy lifestyle habits
* internet access

Exclusion Criteria:

* pregnancy
* diabetes
* heart failure
* coronary artery disease
* kidney disease
* hepatic disease
* cancer
* phenylketonuria
* celiac disease
* food allergies
* bariatric surgery history
* participation in any other weight loss program

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1276 (Actual)
Dates: Start 2017-09-24 (Actual); Primary Completion 2018-04-23 (Actual); Study Completion 2018-04-23 (Actual)

PRIMARY OUTCOMES:
mean weight difference | 24 weeks
  self-reported mean weight difference of 4kg between experimental and control groups

SECONDARY OUTCOMES:
Mean body mass index difference | 24 weeks
  Body mass index difference between experimental and control groups
Daily fruit and vegetables consumption difference | 24 weeks
  Number of daily portions of fruit and vegetables intake difference between experimental and control groups
Sugar-added liquids consumption difference | 24 weeks
  Mean difference in weekly consumption of sugar-added liquids in mL between experimental and control groups
Physical activity classification change | 24 weeks
  Change physical activity level as measured by the International Physical Activity Questionnaire IPAQ

OTHER OUTCOMES:
Quality of life change | 24 weeks
  Quality of life as measured by SF-36 change between control and intervention groups

CONTACTS AND LOCATIONS:
Overall Officials: Alline Maria R Beleigoli, PhD, Principal Investigator — Federal University of Minas Gerais; Andre Q Andrade, PhD, Principal Investigator — University of South Australia; Antonio L Ribeiro, PhD, Principal Investigator — Federal University of Minas Gerais; Maria de Fatima H Diniz, PhD, Study Director — Federal University of Minas Gerais; Roberta S Alvares, MSc, Study Chair — Federal University of Minas Gerais; Leonardo Q Andrade, BSc, Study Chair — Cybergia Tecnologia em Saúde; Tiago M Sizenando, BSc, Study Chair — Cybergia Tecnologia em Saúde
Locations (1):
- Federal University of Minas Gerais, Belo Horizonte, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wadden TA, Butryn ML, Hong PS, Tsai AG. Behavioral treatment of obesity in patients encountered in primary care settings: a systematic review. JAMA. 2014 Nov 5;312(17):1779-91. doi: 10.1001/jama.2014.14173. PMID 25369490
- [Background] Collins CE, Morgan PJ, Jones P, Fletcher K, Martin J, Aguiar EJ, Lucas A, Neve MJ, Callister R. A 12-week commercial web-based weight-loss program for overweight and obese adults: randomized controlled trial comparing basic versus enhanced features. J Med Internet Res. 2012 Apr 25;14(2):e57. doi: 10.2196/jmir.1980. PMID 22555246
- [Background] Hutchesson MJ, Rollo ME, Krukowski R, Ells L, Harvey J, Morgan PJ, Callister R, Plotnikoff R, Collins CE. eHealth interventions for the prevention and treatment of overweight and obesity in adults: a systematic review with meta-analysis. Obes Rev. 2015 May;16(5):376-92. doi: 10.1111/obr.12268. Epub 2015 Mar 5. PMID 25753009
- [Derived] Andrade AQ, Beleigoli A, Diniz MF, Ribeiro AL. Influence of Baseline User Characteristics and Early Use Patterns (24-Hour) on Long-Term Adherence and Effectiveness of a Web-Based Weight Loss Randomized Controlled Trial: Latent Profile Analysis. J Med Internet Res. 2021 Jun 3;23(6):e26421. doi: 10.2196/26421. PMID 34081012
- [Derived] Beleigoli A, Andrade AQ, Diniz MF, Ribeiro AL. Personalized Web-Based Weight Loss Behavior Change Program With and Without Dietitian Online Coaching for Adults With Overweight and Obesity: Randomized Controlled Trial. J Med Internet Res. 2020 Nov 5;22(11):e17494. doi: 10.2196/17494. PMID 33151151
- [Derived] Beleigoli AM, Queiroz de Andrade A, Haueisen Diniz MF, Alvares RS, Ribeiro AL. Online platform for healthy weight loss in adults with overweight and obesity - the "POEmaS" project: a randomized controlled trial. BMC Public Health. 2018 Aug 1;18(1):945. doi: 10.1186/s12889-018-5882-y. PMID 30068393

DOCUMENTS (2):
  • Study Protocol (2018-02-09): https://cdn.clinicaltrials.gov/large-docs/45/NCT03435445/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-09): https://cdn.clinicaltrials.gov/large-docs/45/NCT03435445/SAP_001.pdf